CLINICAL TRIAL: NCT03470493
Title: Comparison of the ApneaLink Air Home Sleep Testing Device to Polysomnography
Brief Title: ApneaLink Air Home Sleep Testing (HST) Device Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SLP-17-10-01
Record Dates: First submitted 2018-02-28; First posted 2018-03-20 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-04

CONDITIONS: Sleep-disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants (Experimental): ApneaLink Air
  Interventions: Diagnostic Test: ApneaLink Air

INTERVENTIONS:
Diagnostic Test: ApneaLink Air — ApneaLink Air to be used on each participant undergoing PSG

SUMMARY:
This study compares the diagnostic capability of a home sleep apnea testing device to polysomnography.

DETAILED DESCRIPTION:
The current gold standard for sleep disordered breathing (SDB) diagnosis is in-laboratory polysomnography (PSG). A barrier of acceptance of Home Sleep Apnea Testing (HSAT) devices as a diagnostic test is their inability to accurately measure total sleep time (TST). A novel algorithm developed by ResMed, Ltd. allows the AL device to accurately calculate TST, however, this algorithm has not yet been validated.

The ApneaLink Air (AL) device is a type III HSAT device. The device is capable of recording up to four channels of data including: flow and snore via a nasal cannula attached to a pressure transducer, a respiratory effort belt, a pulse oximeter to measure pulse and oxygen saturation, and an actigraphy monitor to measure TST along with flow. The AL device has been validated against PSG for AHI, and Cheyne-Stoke respiration detection . Further validation of the effort belt is necessary to determine the accuracy of the AL ability to differentiate between obstructive and central apneic events.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 years of age or older
* Participant is willing to provide informed consent
* Participant is willing to participate in all study related procedures

Exclusion Criteria:

* Unable to cease positive airway pressure (PAP) therapy during PSG (if currently using)
* Requires use of oxygen therapy during sleep
* Diagnosis of uncontrolled clinically relevant sleep disorder (e.g., untreated insomnia or restless leg syndrome)
* Pregnant
* Participant is unsuitable to participate in the study in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berry, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants
Started | 130
Met Primary Endpoint | 80
Completed | 130
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included participants that were considered eligible for the primary endpoint analysis.
Arm/Group | Participants
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 74
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 80
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.1 (8.9)
Current PAP therapy user [Count of Participants; unit: Participants] | 30
Current oxygen user [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Sensitivity of Apnealink (AL) Compared With Polysomnography (PSG)
Description: The Respiratory Event Index (REI) provided by the AL will be compared with the REI provided by the PSG test. REI will be scored according to American Academy of Sleep Medicine (AASM) 2012 guidelines.
  The REI provided by the AL for each participant is divided by the REI provided by the PSG for the same participant to get the diagnostic sensitivity of the Apnealink.
Time Frame: Day 1
Population: Only participants with a respiratory event index (REI) ≥ 5 events per hour according to AL were included in this analysis.
Measure: Number (97.5% Confidence Interval); unit: percent of agreement between AL and PSG
Arm/Group | Participants
Number analyzed (Participants) | 80
percent of agreement between AL and PSG | 91.5 [82.8 to 100]

2. Secondary Outcome: Diagnostic Sensitivity of Apnealink (AL) Compared With Polysomnography (PSG) to Identify Obstructive Events
Description: Total number of Obstructive events reported by the ApneaLink (AL) compared with total number of Obstructive Events reported by polysomnography (PSG). The Obstructive events of the AL are divided by the Obstructive events of the PSG to get the diagnostic sensitivity. This is then compared with the threshold of 0.825
Time Frame: Day 1
Population: Only participants with a respiratory event index (REI) ≥ 5 events per hour according to Apnealink were included in this analysis.
Measure: Number; unit: Weighted Kappa statistic
Arm/Group | Participants
Number analyzed (Participants) | 80
Weighted Kappa statistic | 0.61

3. Secondary Outcome: Diagnostic Sensitivity of the AL to Determine Central Events Compared With PSG
Description: Total number of Central events reported by the ApneaLink (AL) compared with total number of Central Events reported by polysomnography (PSG). The Central events of the AL are divided by the Central events of the PSG to get the diagnostic sensitivity. This is then compared with the threshold of 0.825
Time Frame: Day 1
Population: Only those with an REI over to equal to 5 were included in this analysis
Measure: Number; unit: Weighted Kappa statistic
Arm/Group | Participants
Number analyzed (Participants) | 80
Weighted Kappa statistic | 0.48

4. Secondary Outcome: Positive Likelihood Ratio of Apnealink Air
Description: The positive likelihood ratio (the estimated sensitivity divided by 1 minus the estimated specificity) was calculated along with the associated one-sided 97.5% confidence interval. The positive likelihood ratio was compared with the threshold of 5 (AASM criteria for out-of-center testing devices12) using a Wald test.
Time Frame: Day 1
Population: Only participants with an REI above or equal to 5 were included in this analysis
Measure: Mean (97.5% Confidence Interval); unit: Likelihood Ratio
Arm/Group | Participants
Number analyzed (Participants) | 80
Likelihood Ratio | 3.7 [1.1 to 4.7]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT03470493/Prot_SAP_000.pdf